CLINICAL TRIAL: NCT02186262
Title: Rotating Frame Relaxation and Diffusion Weighted Imaging of Human Gliomas
Acronym: RODIG
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Heikki Minn, Professor, Turku University Hospital
Other Study IDs: 1234
Record Dates: First submitted 2014-07-04; First posted 2014-07-10 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Low Grade Glioma; Malignant Glioma
Keywords: Glioma; MRI; Rotating frame relaxation; DWI; treatment response
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, frozen tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary gliomas, Recurrent gliomas

SUMMARY:
Grading of gliomas is of significant clinical importance since the prognosis as well as the treatment of choice are distinct in low-grade and high-grade gliomas. With standard MRI modalities, however, a reliable distinction is often impossible. Moreover, the gold standard for glioma grading by histopathology may also have limitations due to unrepresentative tumor samples. Therefore, more advanced MRI techniques are urgently needed that would have higher sensitivity and specificity in the definition of tumor type, grade and extent.

Assessment of radiologic response for high-grade gliomas utilizes the updated RANO criteria 12 weeks after completion of chemoradiotherapy. However, there is an urgent need to identify nonresponding patients earlier, preferentially midtreatment in order to consider alternative treatment strategies. Imaging biomarkers, such as diffusion weighted MR imaging (DWI), have provided promising results in assessing early treatment response. Furthermore, a serum biomarker with diagnostic value could improve tumor follow-up and clinical management of gliomas.

The aim of our study is to develop novel imaging protocols suitable for the magnetic resonance imaging (MRI) of glioma using advanced MRI techniques such as rotating frame imaging, novel DWI acquisition and post-processing methods We also study the correlation between advanced MRI parameters and histopathology of the tumor specimen. In addition, early treatment response is assessed with advanced MRI parameters at 3 week and 10 week after initiation of radiotherapy. Finally, our objective is to study the association between serum biomarkers and corresponding MRI with potential tumor progression.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 80 years old
* Language spoken: Finnish or Swedish
* Performance status: Karnofsky score 70 or better or WHO performance status 2 or better
* Supratentorial primary malignant glioma (the diagnosis is based on radiological and clinical grounds)
* Supratentorial recurrent glioma based on MRI and/or [11C]methionine PET imaging
* Patient is scheduled to either surgery or stereotactic biopsy
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethical Committee (EC) approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* Prior medical history: Patient must have no history of serious cardiovascular, liver or kidney disease
* Any psychiatric condition that compromises the subject's ability to participate in the study
* Infections: Patient must not have an uncontrolled serious infection
* No contraindications for MRI (cardiac pacemaker, intracranial clips etc)
* Patient must not have claustrophobia with serious symptoms
* Pregnant or lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a brain tumor scheduled for a surgical resection at the Turku University Hospital, Finland.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-03; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Rotating frame relaxation and diffusion weighted MR parameters in the tumor and surrounding area | Prior to surgical resection
  Different MR relaxation parameters (T1rho-adiabatic,T1rho-cw T2rho-adiabatic,... ) and diffusion values (ADCm, ADCk, K, f, Df, Ds,...) will be measured in the tumor and surrounding area. The quantitative values will be correlated with cancer aggressiveness and tissue bio-markers. Furthermore, tumor volume will be estimated using different quantitative values.

SECONDARY OUTCOMES:
Changes in rotating frame relaxation and diffusion weighted MR parameters in the residual tumor during therapy | Before, after 3 weeks, and after 10 weeks of the beginning of radiotherapy, and 12 weeks after completion of radiotherapy
  Change in the different MR relaxation parameters (T1rho-adaibatic,T1rho-cw T2rho-adiabatic,... ) and diffusion values (ADCm, ADCk, K, f, Df, Ds,...) during tumor therapy will be estimated from repeated MR examinations performed before, after 3 weeks, and after 10 weeks of the beginning of radiotherapy, and 12 weeks after completion of radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Heikki R Minn, Professor, Principal Investigator — Turku University Hospital, Department of Oncology and Radiotherapy
Locations (1):
- Turku University Hospital, Turku, Finland